CLINICAL TRIAL: NCT06021262
Title: Assessment of the Prognostic Value of Nerve Damage Biomarkers in Acute and Chronic Organophosphate Toxicity
Brief Title: Assessment of Nerve Damage Biomarkers in Acute and Chronic Organophosphate Toxicity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed El-Yazbi, Professor, Alexandria University
Other Study IDs: 0107603
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Neuroinflammatory Response; Nerve Injury; Nerve Damage; Neurotoxicity; Nerve Degeneration; Genotoxicity
Keywords: organophosphates; neuroinflammatory biomarkers; metabolomic and proteomic analysis; oxidative stress biomarkers; nerve damage; acute and chronic toxicity; neuroinflammation; inflammatory response; pesticides; acetyl choline esterase enzyme inhibition
MeSH Terms: conditions — Neurotoxicity Syndromes; Nerve Degeneration; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum samples separated from blood samples taken from all study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: healthy individuals without previous acute or chronic exposure to organophosphates
- chronic exposure group: patients with chronic occupational or environmental exposure to organophosphates
  Interventions: Other: exposure to organophosphates
- acute exposure group: patients with acute exposure to organophosphates in accidental or suicidal settings
  Interventions: Other: exposure to organophosphates

INTERVENTIONS:
Other: exposure to organophosphates — organophosphates are esters of phosphoric acids or Thio phosphoric acids that exist in pesticides, where patients can be chronically or acutely exposed to such compounds.
  Groups: acute exposure group; chronic exposure group

SUMMARY:
The aim of this observational study is to answer the following questions in individuals with acute and chronic exposure to organophosphates. The main questions to be addressed are

1. What are the prognostic values of neuroinflammatory markers?
2. What are the genotoxic effects of organophosphates?
3. what are the changes occurring in the levels of traditional oxidative stress and inflammatory markers?

DETAILED DESCRIPTION:
This is a cross-sectional study that aims to assess the possible prognostic value of markers of neuroinflammation and nerve damage in patients with acute and chronic exposure to organophosphate pesticides by conducting a full proteomic and metabolomic profile. The possible genotoxic effect of common organophosphate pesticides will be studied as well. This will be conducted in parallel to the assessment of traditional markers of inflammation and oxidative stress. The target populations are patients with acute and chronic exposure to organophosphates with a total estimated number of 90 including individuals assigned to the control group with matched age and gender.

ELIGIBILITY:
Inclusion Criteria:

* For the control group: healthy individuals without previous exposure to organophosphates, with the specified age limits.
* For the acute exposure group: patients with acute exposure to organophosphates, with the specified age limits
* For the chronic exposure group: patients with chronic exposure to organophosphates, with the specified age limits

No restrictions on comorbidities in the three groups except those mentioned under Exclusion Criteria

Exclusion Criteria:

* Pediatric patients.
* Patients with neurological diseases (Parkinsonism, epilepsy, Alzheimer's disease, etc.)
* Patients who does not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Acute exposure patients will be recruited from the Poison Center and Emergency Department of Alexandria Main University Hospital.
  * Chronic exposure patients will be recruited from farm field workers with a confirmed history of repeated occupational exposure to organophosphate pesticides.
  * Control subjects will be recruited from city dwellers without any medical conditions (healthy subjects) with comparable age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Identification of neuroinflammatory biomarker | 1.5 years
  The biomarker should correlate with nerve injury
Identification of the mechanism of neuroinflammation | 1.5 years
  To detect the possible pathways involved in initiation of systemic inflammation rather than inhibition of choline esterase enzyme. As well as, studying the possible relation of these identified mechanisms with neuronal inflammation and damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

REFERENCES:
- [Background] Syed S, Gurcoo SA, Farooqui AK, Nisa W, Sofi K, Wani TM. Is the World Health Organization-recommended dose of pralidoxime effective in the treatment of organophosphorus poisoning? A randomized, double-blinded and placebo-controlled trial. Saudi J Anaesth. 2015 Jan;9(1):49-54. doi: 10.4103/1658-354X.146306. PMID 25558199
- [Background] Tallat S, Hussien R, Mohamed RH, Abd El Wahab MB, Mahmoud M. Caspases as prognostic markers and mortality predictors in acute organophosphorus poisoning. J Genet Eng Biotechnol. 2020 Apr 13;18(1):10. doi: 10.1186/s43141-020-00024-y. PMID 32281011
- [Background] Rahimi R, Nikfar S, Abdollahi M. Increased morbidity and mortality in acute human organophosphate-poisoned patients treated by oximes: a meta-analysis of clinical trials. Hum Exp Toxicol. 2006 Mar;25(3):157-62. doi: 10.1191/0960327106ht602oa. PMID 16634335
- [Background] Caba IC, Streanga V, Dobrin ME, Jitareanu C, Jitareanu A, Profire BS, Apotrosoaei M, Focsa AV, Caba B, Agoroaei L. Clinical Assessment of Acute Organophosphorus Pesticide Poisoning in Pediatric Patients Admitted to the Toxicology Emergency Department. Toxics. 2022 Oct 2;10(10):582. doi: 10.3390/toxics10100582. PMID 36287862
- [Background] Naughton SX, Terry AV Jr. Neurotoxicity in acute and repeated organophosphate exposure. Toxicology. 2018 Sep 1;408:101-112. doi: 10.1016/j.tox.2018.08.011. Epub 2018 Aug 23. PMID 30144465
- [Background] Lionetto MG, Caricato R, Calisi A, Giordano ME, Schettino T. Acetylcholinesterase as a biomarker in environmental and occupational medicine: new insights and future perspectives. Biomed Res Int. 2013;2013:321213. doi: 10.1155/2013/321213. Epub 2013 Jul 11. PMID 23936791
- [Background] Therkorn J, Drewry DG, Tiburzi O, Astatke M, Young C, Rainwater-Lovett K. Review of Biomarkers and Analytical Methods for Organophosphate Pesticides and Applicability to Nerve Agents. Mil Med. 2020 Mar 2;185(3-4):e414-e421. doi: 10.1093/milmed/usz441. PMID 32077949
- [Background] Kobeissy F, Kobaisi A, Peng W, Barsa C, Goli M, Sibahi A, El Hayek S, Abdelhady S, Ali Haidar M, Sabra M, Oresic M, Logroscino G, Mondello S, Eid AH, Mechref Y. Glycomic and Glycoproteomic Techniques in Neurodegenerative Disorders and Neurotrauma: Towards Personalized Markers. Cells. 2022 Feb 8;11(3):581. doi: 10.3390/cells11030581. PMID 35159390
- [Background] Salvi RM, Lara DR, Ghisolfi ES, Portela LV, Dias RD, Souza DO. Neuropsychiatric evaluation in subjects chronically exposed to organophosphate pesticides. Toxicol Sci. 2003 Apr;72(2):267-71. doi: 10.1093/toxsci/kfg034. PMID 12660361

DOCUMENTS (1):
  • Study Protocol (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT06021262/Prot_000.pdf